CLINICAL TRIAL: NCT03866720
Title: Isolating & Exploiting the Mechanisms That Link Breakfast to Human Health - Acute
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Responsible Party: Principal Investigator, James Betts, Professor James Betts, University of Bath
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: DC-A
Record Dates: First submitted 2019-03-05; First posted 2019-03-07 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Postprandial Metabolism; Appetite

STUDY DESIGN:
Intervention Model Description: Participants will complete 3 breakfast feeding trials in a randomised order:
  Typical high carbohydrate breakfast followed by an ad libitum lunch. Whey protein enriched carbohydrate followed by an ad libitum lunch. Extended morning fast followed by an ad libitum lunch.
Who Masked: Participant
Masking Description: Where applicable (i.e. the two breakfast feeding trials) participants will be blinded to the breakfast that they receive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Carbohydrate rich breakfast (Active Comparator): Participants will consume a porridge breakfast that is considered in line with typical carbohydrate consumption for this meal.
  Interventions: Other: Carbohydrate rich breakfast
- Whey protein enriched breakfast (Experimental): Participants will consume a porridge breakfast that is considered in line with typical carbohydrate consumption for this meal.
  Interventions: Dietary Supplement: Whey protein enriched breakfast
- Extended morning fast (No Intervention): Participants will extend their overnight fast until the ad libitum lunch is provided.

INTERVENTIONS:
Other: Carbohydrate rich breakfast — A porridge breakfast meal fed at a carbohydrate delivery rate of 7.3 mg/kJ of each participants resting metabolic rate.
  Arms: Carbohydrate rich breakfast
Dietary Supplement: Whey protein enriched breakfast — A porridge breakfast meal in which 15 grams of whey protein is substituted in place of carbohydrate and a small portion of fat.
  Arms: Whey protein enriched breakfast

SUMMARY:
Following the establishment of causal links between breakfast consumption, the individual components of energy balance, and health it is now important to examine and target the underlying biological mechanisms involved to maximise potential health benefits.

To begin investigating the outlined mechanisms healthy, non-obese participants will be recruited to take part in phase I (acute crossover design) of a wider project.

DETAILED DESCRIPTION:
Causal links between breakfast consumption, the individual components of energy balance, and health have recently been established and it is now important to examine and target the underlying biological mechanisms involved to maximised potential health benefits.

Specifically, the substitution of a portion of carbohydrate for protein at breakfast may enhance the potential health benefits of breakfast through targeting distinct mechanistic pathways. Broadly, introducing a greater protein load at breakfast increases insulin secretion and delays gastric emptying, thereby eliciting a potentiated insulin response. In turn this may therefore improve glucose tolerance during a subsequent meal. Additionally, maintenance of euglycaemia following breakfast consumption, coupled with the thermic effect of feeding protein may accentuate the elevated energy expenditure following breakfast observed in previous studies. Finally, both the physical and chemical properties of protein exert a marked satiating effect. Collectively, these mechanisms could interact to maximise the net impact of breakfast on energy balance and associated health outcomes. However, whilst the evidence indicates obvious benefits of feeding a higher protein dose at breakfast, relatively little research has focused on the response to protein over multiple meals/days. Furthermore, and importantly, the mechanisms involved in the second-meal phenomenon and the potential for initial meals of varied composition to target these mechanisms have never been systematically investigated.

To begin investigating the outlined mechanisms healthy, non-obese participants will be recruited to take part a randomised crossover trial that will contrast the acute metabolic responses to a protein-enriched breakfast, with a carbohydrate rich breakfast, and the total omission of breakfast.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 18.5-29.9 kg∙m-2
* Age 18-65 years
* Able and willing to provide informed consent and safely comply with study procedures
* Females to maintain record of regular menstrual cycle phase or contraceptive use
* No anticipated changes in diet/physical activity during the study (e.g. holidays or diet plans)
* Inclusive to all breakfast habits (e.g. regular skipper / consumer)

Exclusion Criteria:

* Any reported condition or behaviour deemed either to pose undue personal risk to the participant or introduce bias
* Any diagnosed metabolic disease (e.g. type 1 or type 2 diabetes)
* Any reported use of substances which may pose undue personal risk to the participants or introduce bias into the experiment (e.g. smoking/substance abuse)
* Lifestyle not conforming to standard sleep-wake cycle (e.g. shift worker)
* Any reported recent (<6 months) change in body mass (± 3%)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2021-02-17 (Actual); Study Completion 2021-02-17 (Actual)

PRIMARY OUTCOMES:
Postprandial glycaemia following breakfast | Plasma glucose time course data over 3 hours following breakfast
  The postprandial time course response of plasma glucose to each breakfast meal
Postprandial insulinaemia following breakfast | Plasma insulin time course data over 3 hours following breakfast
  The postprandial time course response of plasma insulin to each breakfast meal
Postprandial glycaemia following ad libitum lunch | Plasma glucose time course data over 2 hours following lunch
  The postprandial time course response of Plasma glucose to the ad libitum lunch following each type of breakfast
Postprandial insulinaemia following ad libitum lunch | Plasma insulin time course data over 2 hours following lunch
  The postprandial time course response of plasma insulin to the ad libitum lunch following each type of breakfast

SECONDARY OUTCOMES:
Postprandial incretin hormone response following breakfast | Plasma insulin time course data over 3 hours following breakfast
  The postprandial time course response of plasma incretin hormones (e.g. GLP-1 & GIP) to the each breakfast.
Postprandial incretin hormone response following ad libitum lunch | Plasma incretin time course data over 3 hours following breakfast
  The postprandial time course response of plasma incretin hormones (e.g. GLP-1 & GIP) to the ad libitum lunch following each type of breakfast
Subjective appetite ratings following breakfast | For 3 hours following each breakfast
  Ratings of appetite provided on subjective appetite scales following each type of breakfast. On a scale of 0-100mm with 0 typically being associated with lower subjective ratings and 100 being associated with higher subjective ratings.
Subjective appetite ratings following ad libitum lunch | For 3 hours following the ad libitum lunch
  Ratings of appetite provided on subjective appetite scales following ad libitum lunch. On a scale of 0-100mm with 0 typically being associated with lower subjective ratings and 100 being associated with higher subjective ratings.
Fuel oxidation following breakfast | For 3 hours following breakfast
  Fat and carbohydrate oxidation following each type of breakfast
Fuel oxidation following ad libitum lunch | For 2 hours following the ad libitum lunch
  Fat and carbohydrate oxidation following ad libitum lunch

CONTACTS AND LOCATIONS:
Overall Officials: Harry A Smith, MSci, Principal Investigator — University of Bath; James A Betts, PhD, Principal Investigator — University of Bath
Locations (1):
- University of Bath, Bath, Somerset, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chowdhury EA, Richardson JD, Tsintzas K, Thompson D, Betts JA. Carbohydrate-rich breakfast attenuates glycaemic, insulinaemic and ghrelin response to ad libitum lunch relative to morning fasting in lean adults. Br J Nutr. 2015 Jul 14;114(1):98-107. doi: 10.1017/S0007114515001506. Epub 2015 May 25. PMID 26004166
- [Background] Park YM, Heden TD, Liu Y, Nyhoff LM, Thyfault JP, Leidy HJ, Kanaley JA. A high-protein breakfast induces greater insulin and glucose-dependent insulinotropic peptide responses to a subsequent lunch meal in individuals with type 2 diabetes. J Nutr. 2015 Mar;145(3):452-8. doi: 10.3945/jn.114.202549. Epub 2014 Dec 24. PMID 25733459
- [Background] Bray GA, Redman LM, de Jonge L, Covington J, Rood J, Brock C, Mancuso S, Martin CK, Smith SR. Effect of protein overfeeding on energy expenditure measured in a metabolic chamber. Am J Clin Nutr. 2015 Mar;101(3):496-505. doi: 10.3945/ajcn.114.091769. Epub 2015 Jan 14. PMID 25733634
- [Background] Leidy HJ, Ortinau LC, Douglas SM, Hoertel HA. Beneficial effects of a higher-protein breakfast on the appetitive, hormonal, and neural signals controlling energy intake regulation in overweight/obese, "breakfast-skipping," late-adolescent girls. Am J Clin Nutr. 2013 Apr;97(4):677-88. doi: 10.3945/ajcn.112.053116. Epub 2013 Feb 27. PMID 23446906
- [Derived] Smith HA, Watkins JD, Walhin JP, Gonzalez JT, Thompson D, Betts JA. Whey Protein-Enriched and Carbohydrate-Rich Breakfasts Attenuate Insulinemic Responses to an ad libitum Lunch Relative to Extended Morning Fasting: A Randomized Crossover Trial. J Nutr. 2023 Oct;153(10):2842-2853. doi: 10.1016/j.tjnut.2023.08.008. Epub 2023 Aug 7. PMID 37557957